CLINICAL TRIAL: NCT03884842
Title: A Two-arm, Placebo-controlled Randomized Clinical Trial to Evaluate the Effect of Dupilumab on Airway Hyper-responsiveness and Ventilation Heterogeneity in Patients With Asthma With a "T2 Immune Signature"
Brief Title: Dupilumab on Airway Hyper-responsiveness and Ventilation Heterogeneity in Patients With Asthma.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11963
Record Dates: First submitted 2019-03-18; First posted 2019-03-21 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Asthma
Keywords: Airway hyperresponsivness; Ventilation heterogeneity; Hyperpolarized Xenon-129; Sputum eosinophils
MeSH Terms: conditions — Asthma | interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dupilumab (Active Comparator): Dupilumab 300 mg subcutaneously (SC) every 2 weeks as an investigational drug. For those randomized to dupilumab, a loading dose of 600 mg will be given only at randomization/Visit 2.
  Sterile dupilumab of will be provided in 150 mg/mL in glass prefilled syringes (2.25 mL total volume) to deliver 300 mg in 2 mL.
  Interventions: Biological: Dupilumab/Dupixent
- matched placebo (Placebo Comparator): Sterile placebo for dupilumab will be provided in identically matched glass prefilled syringes to deliver 2 mL.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Dupilumab/Dupixent — a monoclonal antibody designed for the treatment asthma and atopic dermatitis.
  Arms: dupilumab
Biological: Placebo — Matched placebo
  Arms: matched placebo

SUMMARY:
In asthmatics with airway hyperresponsiveness and a "T2 immune signature" (type 2), Dupilumab will suppress airway hyperresponsiveness (assessed by methacholine PC20 ≤ 4 mg/mL (PC20: provocative concentration causing a 20% fall in FEV1) OR ≥15% decreased in forced expired volume in 1 second (FEV1) during saline inhalation for sputum induction OR ≥25% improvement in FEV1 after bronchodilator) and airway eosinophilia (assessed by sputum eosinophils) and this will be associated with greater asthma control and improved ventilation heterogeneity.

DETAILED DESCRIPTION:
Along with these features of eosinophil recruitment, degranulation and autoantibody generation, that are partly dependent on (interleukin-4) IL-4 and (interleukin-13) IL-13 signalling, two additional characteristic features of asthma ie airway hyperresponsiveness and mucus hypersecretion are also determined by IL-13 biology. Neither of these important features have been investigated in any clinical trials of anti-IL-13 molecules. Accurate endotyping to identify patients in whom IL-13 mediated biology is the dominant pathobiology of asthma (selecting patients with significant airway hyperresponsiveness and mucus secretion) may elicit greater clinical effect. Taken together, we propose to investigate the effects of Dupilumab on airway hyperresponsiveness, on airway eosinophilia and mucus biology and their relation to airway structure and function (ventilation heterogeneity), and airway autoimmune responses.

To satisfy the proposed objective we will evaluate well-established outcome measures of airway hyperresponsiveness (provocation concentration of methacholine causing a 20% fall in FEV1 (PC20), type 2 inflammation (sputum eosinophils, blood eosinophils and exhaled nitric oxide (eNO)) and mucus biology.

ELIGIBILITY:
Inclusion Criteria:

* General

  1. Able and willing to provide written informed consent.
  2. Able and willing to comply with the study protocol.
  3. Males and females ≥ 18 years of age.

     Asthma-related
  4. Asthma diagnosed by a respiratory physician ≥ 12 months prior to study enrolment based on the Global Initiative for Asthma (GINA) 2014 guidelines.
  5. ACQ > 1 during the screening period.
  6. Airway hyperresponsiveness (methacholine PC20 ≤ 4 mg/mL OR ≥15% decreased in FEV1 during saline inhalation for sputum induction OR ≥25% improvement in FEV1 after bronchodilator) during the screening period.
  7. Fraction of exhaled nitric oxide (FeNO) >25 ppb and either ≥3% sputum eosinophils (preferred) OR blood eos ≥300/µL during the screening period.
  8. Inhaled corticosteroids (ICS) dose ≥500 mcg of fluticasone equivalent/day. Patients on prednisone would not be excluded as long as they meet the rest of the inclusion criteria.

Exclusion Criteria:

* Patients who meet any of the following criteria will be excluded from study entry:

Prior Medical Conditions and Treatment History

1. Acute or chronic parasitic, bacterial, fungal or viral infections that required, or currently requires, hospitalization or antimicrobial treatment during the last four weeks.
2. Acute asthma exacerbation event treated with increased doses of oral, or any dose of intramuscular (IM) or intravenous (IV) corticosteroids within six weeks prior to screening.
3. Other relevant pulmonary diseases (e.g. chronic obstructive pulmonary disease, idiopathic pulmonary fibrosis, cystic fibrosis, pulmonary arterial hypertension, tuberculosis) requiring treatment within 12 months prior to screening.
4. Alcohol or substance abuse within 12 months prior to screening.
5. Current smoker defined as having smoked at least one cigarette (or pipe, cigar, or marijuana) per day for ≥ 30 days within the three months prior to screening.
6. Ex-smokers with ≥ 10 pack-year smoking history.
7. Treatment with anti-IgE (immunoglobulin E), anti-IL-4, anti-IL-5 (interleukin-5), or anti-IL-13 targeted therapy currently or within three months prior to screening.
8. ACQ > 3.0

   MRI (Magnetic Resonance Imaging )Related
9. Patient has an implanted mechanically, electrically or magnetically activated device or any metal in their body which cannot be removed, including but not limited to pacemakers, neurostimulators, biostimulators, implanted insulin pumps, aneurysm clips, bioprosthesis, artificial limb, metallic fragment or foreign body, shunt, surgical staples (including clips or metallic sutures and/or ear implants) (at the discretion of the MRI Technologist).
10. In the investigator's opinion, subject suffers from any physical, psychological or other condition(s) that might prevent performance of the MRI, such as severe claustrophobia.

    General
11. Participation in any clinical trial of an investigational agent or procedure within six months prior to screening or during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-10-12 (Actual); Study Completion 2023-01-17 (Actual)

PRIMARY OUTCOMES:
Proportion of patients that achieve at least one doubling dose improvement in PC20 methacholine and/or a 50% reduction in FEV1 reversibility after bronchodilator. | Between screening (week -4) and week 16.
  For patients that can undergo a methacholine challenge, one doubling dose improvement in PC20 methacholine. For those that cannot undergo a methacholine challenge a 50% reduction in FEV1 reversibility.

SECONDARY OUTCOMES:
Change in geometric mean PC20 methacholine. | Between screening (week -4) and week 16.
  Change in PC20 between screening and week 16.
Change in FEV1 reversibility. | Between randomization (week 0) and week 16.
  Change in FEV1 % reversibility (pre/post bronchodilator) between randomization and end of treatment.
Change in sputum eosinophil percentage (%) | Between randomization (week 0) and week 16.
  Change in sputum eosinophil percentage between randomization and end of treatment
Change in blood eosinophil count | Between randomization (week 0) and week 16.
  Change in blood eosinophil count levels between randomization and end of treatment
Change in fraction of exhaled nitric oxide (FeNO) | Between randomization (week 0) and week 16.
  Change in FeNO values parts per billion (ppb) from randomization and end of treatment.
Change in FEV1 (pre-bronchodilator) | Between randomization (week 0) and week 16.
  Change in pre-bronchodilator FEV1 values (in litres) between randomization and end of treatment.
Change in Asthma Control Questionnaire-5 (ACQ-5) | Between randomization (week 0) and week 16.
  Change in ACQ scores between randomization and end of treatment.
Change in Asthma Control Questionnaire-5 (AQLQ) | Between randomization (week 0) and week 16.
  Change in AQLQ scores between randomization and end of treatment.
Change in Asthma Control Test (ACT) | Between randomization (week 0) and week 16.
  Change in ACT scores between randomization and end of treatment.

OTHER OUTCOMES:
Change in MRI ventilation heterogeneity (n=12 in each arm). | Between randomization (week 0) and week 16.
  Change in MRI ventilation heterogeneity seen with administration of Hyperpolarized Xenon-129 inhalation.
Change in CT airway remodeling and airway mucus scores (n=12 in each arm). | Between randomization (week 0) and week 16.
  Changes are evaluated via CT inspiratory/expiratory scans via quantitative software (n=12 in each arm)

CONTACTS AND LOCATIONS:
Overall Officials: Parameswaran Nair, MD, PhD, Principal Investigator — McMaster University
Locations (1):
- Firestone Institute for Respiratory Health, St. Joseph's Healthcare, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wills-Karp M, Luyimbazi J, Xu X, Schofield B, Neben TY, Karp CL, Donaldson DD. Interleukin-13: central mediator of allergic asthma. Science. 1998 Dec 18;282(5397):2258-61. doi: 10.1126/science.282.5397.2258. PMID 9856949
- [Background] Svenningsen S, Kirby M, Starr D, Leary D, Wheatley A, Maksym GN, McCormack DG, Parraga G. Hyperpolarized (3) He and (129) Xe MRI: differences in asthma before bronchodilation. J Magn Reson Imaging. 2013 Dec;38(6):1521-30. doi: 10.1002/jmri.24111. Epub 2013 Apr 15. PMID 23589465
- [Background] Crapo RO, Casaburi R, Coates AL, Enright PL, Hankinson JL, Irvin CG, MacIntyre NR, McKay RT, Wanger JS, Anderson SD, Cockcroft DW, Fish JE, Sterk PJ. Guidelines for methacholine and exercise challenge testing-1999. This official statement of the American Thoracic Society was adopted by the ATS Board of Directors, July 1999. Am J Respir Crit Care Med. 2000 Jan;161(1):309-29. doi: 10.1164/ajrccm.161.1.ats11-99. No abstract available. PMID 10619836
- [Derived] Svenningsen S, Kjarsgaard M, Haider E, Venegas C, Konyer N, Friedlander Y, Nasir N, Boylan C, Kirby M, Nair P. Effects of Dupilumab on Mucus Plugging and Ventilation Defects in Patients with Moderate-to-Severe Asthma: A Randomized, Double-Blind, Placebo-Controlled Trial. Am J Respir Crit Care Med. 2023 Nov 1;208(9):995-997. doi: 10.1164/rccm.202306-1102LE. No abstract available. PMID 37603097